CLINICAL TRIAL: NCT00108628
Title: 7857 Cognitive - Behavioral Treatments for PTSD Sleep Disturbance
Brief Title: Cognitive Behavioral Treatments for Post-traumatic Stress Disorder (PTSD) Sleep Disturbance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN-018-03S
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Imagery; Nightmares; Post-Traumatic Stress Disorder; Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Imagery Rehearsal Therapy
  Interventions: Behavioral: Imagery Rehearsal
- Arm 2 (Active Comparator): Sleep and Nightmare Management
  Interventions: Behavioral: Sleep and Nightmare Management

INTERVENTIONS:
Behavioral: Imagery Rehearsal — IR is a manual-based CBT predicated on the idea that waking mental activity influences nighttime dreams. Veterans examine the content of a recurrent nightmare, use imagery to alter disturbing aspects of the nightmare to promote mastery and control, and rehearse the new dream nightly, before bedtime.
  Arms: Arm 1
Behavioral: Sleep and Nightmare Management — This comparison condition involved psychoeducation about PTSD, sleep and nightmares, progressive muscle relaxation and standard CBT for insomnia. This latter part included education about sleep hygiene (e.g., avoidance of caffeine and alcohol close to bedtime, benefit of regular bed time routines), stimulus control and sleep restriction (i.e., reestablishing a conditioned association between the bed/bedroom and sleep by reducing time spent tossing and turning in bed). Therapists worked with patients to identify problem areas in their sleep habits and to problem-solve about possible treatment targets
  Arms: Arm 2

SUMMARY:
The purpose of this study is to compare the effectiveness of two cognitive behavioral group psychotherapy interventions in controlling the subjective sleep disturbance in veterans with Post-traumatic Stress Disorder.

DETAILED DESCRIPTION:
Repetitive, stereotypical nightmares and insomnia commonly characterize post-traumatic stress disorder (PTSD). Identifying the pathophysiological mechanisms of disrupted sleep in PTSD has therefore assumed considerable clinical importance. We previously reported an increase in rapid eye movement activity (REM activity) during REM sleep (REMS) in Vietnam War combat veterans with PTSD, and this finding can be seen as consistent with the view that most, although not all, dreaming occurs during REMS and the repeated observation that REM activity correlates with the intensity of dream mentation. There is a growing body of evidence that post-traumatic nightmares can respond to psychological treatment interventions. Namely, a cognitive-behavioral technique entitled imagery rehearsal (IR) has been reported to be effective in the treatment of such nightmares in victims of crime and in women who have been sexually assaulted. In a small pilot study, it has also been reported to be effective in the treatment of Vietnam veterans with combat-related PTSD. The two objectives of this proposal are: 1. To compare, in a study with random assignment and a parallel group design, the effectiveness in controlling the subjective sleep disturbance in veterans with PTSD of IR and Sleep and Nightmare Management (SN), a psychological treatment that targets life stressors and problems with sleep hygiene that may exacerbate insomnia and nightmares. 2. In a subset of these subjects, to compare the effectiveness in reducing REM activity of IR and SN.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Vietnam Combat Veteran
* Diagnosis of combat-related PTSD
* Stable psychotropic regimen for a minimum of three months
* Experiences recurrent nightmares

Exclusion Criteria:

* Bipolar disorder, delirium, dementia, amnestic and other cognitive disorders
* Schizophrenia and other psychotic disorders
* Substance abuse or dependence within the last six months
* Untreated medical disorders known to impact sleep

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2004-04; Primary Completion 2008-09 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Ross, MD PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center
Locations (1):
- Philadelphia VA Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Harb GC, Thompson R, Ross RJ, Cook JM. Combat-related PTSD nightmares and imagery rehearsal: nightmare characteristics and relation to treatment outcome. J Trauma Stress. 2012 Oct;25(5):511-8. doi: 10.1002/jts.21748. Epub 2012 Oct 9. PMID 23047646
- [Result] Cook JM, Harb GC, Gehrman PR, Cary MS, Gamble GM, Forbes D, Ross RJ. Imagery rehearsal for posttraumatic nightmares: a randomized controlled trial. J Trauma Stress. 2010 Oct;23(5):553-63. doi: 10.1002/jts.20569. PMID 20839311
- [Result] Cook JM, Thompson R, Harb GC, Ross RJ. Cognitive-behavioral treatment for posttraumatic nightmares: An investigation of predictors of dropout and outcome. Psychological trauma : theory, research, practice and policy. 2013 Nov 1; 5(6):545-553.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ten participants dropped out prior to randomization.
Groups:
- Imagery Rehearsal Therapy: Imagery Rehearsal Therapy
  Imagery Rehearsal: IR is a manual-based CBT predicated on the idea that waking mental activity influences nighttime dreams. Veterans examine the content of a recurrent nightmare, use imagery to alter disturbing aspects of the nightmare to promote mastery and control, and rehearse the new dream nightly, before bedtime.
- Sleep and Nightmare Management: Sleep and Nightmare Management
  Sleep and Nightmare Management: This comparison condition involved psychoeducation about PTSD, sleep and nightmares, progressive muscle relaxation and standard CBT for insomnia. This latter part included education about sleep hygiene (e.g., avoidance of caffeine and alcohol close to bedtime, benefit of regular bed time routines), stimulus control and sleep restriction (i.e., reestablishing a conditioned association between the bed/bedroom and sleep by reducing time spent tossing and turning in bed). Therapists worked with patients to identify problem areas in their sleep habits and to problem-solve about possible treatment targets
Period: Overall Study
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Started | 61 | 63
Received One or More Sessions | 53 | 58
Completed Treatment | 42 | 57
Completed | 41 | 53
Not Completed | 20 | 10
Not completed — Withdrawal by Subject | 17 | 9
Not completed — Lack of Efficacy | 2 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management | Total
Number analyzed (Participants) | 61 | 63 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.79 (3.18) | 59.06 (3.86) | 59.42 (3.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 61 | 63 | 124
Region of Enrollment [Number; unit: participants]
  United States | 61 | 63 | 124

OUTCOME MEASURES:

1. Primary Outcome: Weekly Number of Nightmares
Time Frame: Baseline and 1, 3, and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: weekly nightmares
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Number analyzed (Participants) | 61 | 63
weekly nightmares
  Baseline | 3.95 (2.37) | 3.88 (3.95)
  1 month | 3.28 (2.47) | 3.47 (2.72)
  3 months | 3.61 (2.63) | 3.09 (2.08)
  6 months | 3.20 (2.14) | 3.04 (1.89)

2. Primary Outcome: Weekly Nights With a Nightmare
Time Frame: Baseline and 1, 3, and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: nights/week
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Number analyzed (Participants) | 61 | 63
nights/week
  Baseline | 2.96 (1.39) | 3.00 (1.43)
  1 month | 2.67 (1.64) | 2.78 (1.54)
  3 months | 3.10 (1.70) | 2.55 (1.41)
  6 months | 2.98 (1.69) | 2.68 (1.42)

3. Primary Outcome: Pittsburgh Sleep Quality Index
Description: Total scores range from 0 to 21, with higher values indicating poorer sleep quality. A score greater than 5 distinguishes between poor and good sleepers.
Time Frame: Baseline and 1, 3, and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Number analyzed (Participants) | 61 | 63
units on a scale
  Baseline | 13.40 (3.00) | 12.85 (3.32)
  1 month | 12.09 (4.26) | 11.82 (3.79)
  3 months | 12.57 (3.83) | 11.70 (3.90)
  6 months | 12.06 (4.09) | 12.00 (4.51)

4. Secondary Outcome: Pittsburgh Sleep Quality Index - Addendum
Description: The PSQI-A is a measure of PTSD-related sleep and dream disturbances. Scores can range from 0 to 21, with higher scores reflecting greater sleep problems.
Time Frame: Baseline and 1, 3, and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Number analyzed (Participants) | 61 | 63
units on a scale
  Baseline | 17.51 (4.96) | 17.01 (3.76)
  1 month post-treatment | 16.71 (5.18) | 16.29 (3.91)
  3 months post-treatment | 16.58 (5.56) | 16.36 (4.16)
  6 months post-treatment | 17.35 (5.13) | 17.26 (4.56)

5. Secondary Outcome: Nightmare Effects Survey
Description: This self-report questionnaire assesses psychosocial impairment attributed to nightmares. Eleven self-report questions are rated on a scale of zero to four. The individual scores are summed to produce a total score ranging from 0 to 44 (reported in the Table). Higher scores reflect greater impairment.
Time Frame: Baseline and 1, 3, and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Number analyzed (Participants) | 61 | 63
units on a scale
  Baseline | 26.39 (9.00) | 24.11 (9.99)
  1 month post-treatment | 24.12 (10.43) | 24.66 (9.18)
  3 months post-treatment | 25.28 (10.06) | 24.02 (10.22)
  6 months post-treatment | 25.88 (9.75) | 24.98 (10.14)

6. Secondary Outcome: PTSD Military Checklist
Description: Seventeen items indicating the 17 DSM-IV criteria for PTSD are rated on a 5-point scale, from 1 to 5. Scores range from 17 to 85, with a higher score indicating greater symptom severity.
Time Frame: Baseline and 1, 3, and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Number analyzed (Participants) | 61 | 63
units on a scale
  Baseline | 62.73 (10.18) | 65.06 (9.48)
  1 month post-treatment | 58.83 (13.56) | 60.96 (11.43)
  3 months post-treatment | 60.13 (12.16) | 61.13 (12.00)
  6 months post-treatment | 59.05 (11.87) | 59.64 (12.30)

7. Secondary Outcome: Beck Depression Inventory
Description: Twenty-one items are rated on a 4-point scale. Total scores range from zero to 63, with higher scores indicating more severe depression.
Time Frame: Baseline and 1, 3, and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Number analyzed (Participants) | 61 | 63
units on a scale
  Baseline | 26.85 (11.82) | 23.51 (11.92)
  1 month post-treatment | 24.16 (13.35) | 22.31 (12.76)
  3 months post-treatment | 24.80 (13.14) | 23.76 (12.76)
  6 months post-treatment | 25.02 (13.30) | 23.37 (12.34)

8. Secondary Outcome: SF-36 Physical Component
Description: The Health Assessment Questionnaire Short Form 36 (SF-36) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Scales 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Scores on each scale are summed and averaged (range = 0 "worst"-100 "best").
Time Frame: Baseline and 1, 3, and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Number analyzed (Participants) | 61 | 63
units on a scale
  Baseline | 37.17 (9.21) | 38.53 (9.64)
  1 month post-treatment | 39.48 (10.19) | 36.84 (10.34)
  3 months post-treatment | 37.72 (9.57) | 35.96 (11.97)
  6 months post-treatment | 35.80 (9.64) | 37.21 (11.23)

9. Secondary Outcome: SF-36 Mental Component
Description: The Health Assessment Questionnaire Short Form 36 (SF-36) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Scales 5-8 primarily contribute to the mental component summary score (PCS) of the SF-36. Scores on each scale are summed and averaged (range = 0 "worst"-100 "best").
Time Frame: Baseline and 1, 3, and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Number analyzed (Participants) | 61 | 63
units on a scale
  Baseline | 29.69 (9.08) | 34.52 (12.06)
  1 month post-treatment | 32.33 (10.63) | 32.84 (9.75)
  3 months post-treatment | 30.98 (9.33) | 34.00 (10.35)
  6 months post-treatment | 32.15 (8.99) | 34.78 (10.87)

10. Secondary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: Seventeen questions assess the frequency and intensity of PTSD symptoms. Scores range from zero to 136, with a higher score indicating more severe symptoms.
Time Frame: Baseline and 1 month post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Number analyzed (Participants) | 61 | 63
units on a scale
  Baseline | 81.34 (14.00) | 79.48 (15.27)
  1 month post-treatment | 74.04 (20.36) | 74.85 (19.52)

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were not assessed
Arm/Group | Imagery Rehearsal Therapy | Sleep and Nightmare Management
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/58
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes